CLINICAL TRIAL: NCT06137521
Title: Risk Factors and Outcomes in Patients With Stable Coronary Artery Disease and Coronary Chronic Total Occlusion
Brief Title: Risk Factors and Outcomes in Coronary Chronic Total Occlusion
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RFOCTO
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Total Occlusion; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with good coronary collaterals: Coronary collateral circulation development was graded according to the Rentrop score, grade 2 (partial filling of the epicardial segment by collateral vessels); grade 3 (complete filling of the epicardial artery by collateral vessels) were defined as good coronary collateral circulation.
  Interventions: Procedure: Coronary angiography
- Patients with poor coronary collaterals: Coronary collateral circulation development was graded according to the Rentrop score, grade 0 (no filling of any collateral vessels) and grade 1 (filling of side branches of the artery to be perfused by collateral vessels without visualization of the epicardial segment) were defined as poor coronary collateral circulation.
  Interventions: Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Coronary angiography

SUMMARY:
This study aims to assess the risk factors and evaluate the long-term outcomes of patients with coronary chronic total occlusion (CTO) treated with percutaneous coronary intervention or medical treatment.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is still one of the major contributors to global mortality. CTO is a special lesion type of CAD, defined as complete occlusion of at least one major epicardial coronary artery more than 3 months. Compared to non-CTO patients, those with CTO have worse prognosis. The prognosis of CTO patients is related to many factors including the baseline characteristics, modality of treatment and the degree of coronary collateral formation. Figuring out the factors which can indicate the outcomes of CTO is essential to clinical decision making. In this single center, observational study, we collect patient's clinical characteristics and blood samples to investigate potential factors associated with the development of coronary collateral formation and outcomes in patents with stable coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years; Patients with angina or silent ischemia and documented ischemia; Patients with CTO ≥ 3months

Exclusion Criteria:

* eGFR<15mL/(min·1.73m2); Chronic heart failure with NYHA grade ≥3; Had a history of coronary artery bypass grafting; Had received a percutaneous coronary intervention within the prior 3 months; Malignant tumor or immune system disorders; Pulmonary heart disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease and CTO undergone coronary angiography at Ruijin Hospital, Shanghai, China will be consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The degree of collateral estimated visually by Rentrop score during coronary angiography | Immediate post-angiography
  The degree of coronary collateralization supplying the distal area of the total coronary occlusion was visually graded using the Rentrop scoring system as follows: 0=no visible collaterals; 1=poorly opacified collaterals with faint visualization of the distal vessel; 2=partial filling of the collateral vessels; and 3=complete filling of the collateral vessels. Patients were then classified as poor coronary collaterals (Rentrop scores of 0 and 1) or good coronary collaterals (Rentrop scores of 2 and 3), according to the Rentrop score.
Composite event of all-cause mortality, non-fatal myocardial infarction, heart failure and repeat revascularization | up to 5 years

SECONDARY OUTCOMES:
Event of all-cause mortality | up to 5 years
Event of death from cardiac causes | up to 5 years
Event of heart failure | up to 5 years
The change of left ventricular ejection fraction | 1 year
Events of repeat revascularization | up to 5 years
Event rate of procedural success | Immediate post-PCI
Event of procedural outcomes | 1 month post-angiography or PCI

OTHER OUTCOMES:
The level of serum markers and biochemical indexes which have been reported to closely related to cardiovascular diseases and collateral formation. | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fenghua Ding, PhD, MD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China